CLINICAL TRIAL: NCT01233934
Title: Comparative Study of Two Forms of Topical Dexchlorpheniramine Maleate (Cream Versus Gel) for Insect Bites
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Celso Sustovich, Medical Director
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERP 185v3-10
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Insect Bites
Keywords: Insect bites; Dexchlorpheniramine; Gel; Cream
MeSH Terms: conditions — Insect Bites and Stings | interventions — dexchlorpheniramine; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexchlorpheniramine 1% Cream (Active Comparator)
  Interventions: Drug: Dexchlorpheniramine 1% Cream
- Dexchlorpheniramine 1% Gel (Experimental)
  Interventions: Drug: Dexchlorpheniramine 1% Gel

INTERVENTIONS:
Drug: Dexchlorpheniramine 1% Gel — Small amount applied over the lesion twice a day for 7 days.
  Arms: Dexchlorpheniramine 1% Gel
Drug: Dexchlorpheniramine 1% Cream — Small amount applied over the lesion twice a day for 7 days.
  Arms: Dexchlorpheniramine 1% Cream

SUMMARY:
Insect bite related symptoms (pruritus and papules) are caused by the release of histamine by mast cells in the skin. Topical anti-histaminics can be used to promote relief of these symptoms. Dexchlorpheniramine maleate 1% cream is a topical anti-histaminic formulation approved by ANVISA in Brazil for the relief of skin irritation and allergies, including the ones caused by insect bites. The aim of the present study is to demonstrate non-inferiority of a new pharmacological preparation of dexchlorpheniramine maleate (1% gel) with the standard preparation (1% cream) for the relief of insect bite related symptoms and to demonstrate the safety of both preparations.

ELIGIBILITY:
Inclusion Criteria:

* Presence of papules resulting from insect bites within the last 72 hours;
* Presence of symmetric lesions to compare one side to the other;
* Compliance of the subject to the treatment protocol;
* Agreement with the terms of the informed consent by the participants or their legal guardians when younger than 18 years old.

Exclusion Criteria:

* Pregnancy or risk of pregnancy;
* Lactation;
* Use of topical or systemic anti-inflammatory, anti-histaminics or immunosuppressive drugs within the last 48 hours prior to the study;
* History of atopy or allergic diseases;
* History of allergy of any component of the formulations;
* Other conditions considered by the investigator as reasonable for non-eligibility.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Pruritus Intensity at Insect Bite Site, Evaluated With a 10 Point Visual Analogic Scale (VAS) | 7 days

SECONDARY OUTCOMES:
Composite Clinical Evaluation of Erythema, Pruritus and Papule Formation, Performed by the Investigator Using a 4-point Scale for Each One of the Parameters (Absent, Mild, Moderate, Intense). This Evaluation Constitutes the Insect Bite Score. | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele Ltda., Osasco, São Paulo, Brazil